CLINICAL TRIAL: NCT03532776
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, Placebo- Controlled, Study of Hyloris Developments' Podofilox Topical Gel 0.5% Compared to Allergan's Condylox® Gel 0.5% in Male and Female Patients With External Anogenital Warts.
Brief Title: Comparison Between Podofilox Topical Gel 0.5% and Allergan's Condylox® Gel 0.5% for External Anogenital Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dermax SA (Industry)
Collaborators: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 016-POD-001
Record Dates: First submitted 2018-01-11; First posted 2018-05-22 (Actual); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2019-02

CONDITIONS: External Anogenital Warts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Podofilox Gel 0.5 % (Experimental): Podofilox Gel 0.5% twice a day, three days following by four days of discontinuation, up to four cycles
  Interventions: Drug: Podofilox Gel 0.5%
- Condylox Topical Gel 0.5% (Active Comparator): Condylox Topical Gel 0.5% twice daily, three days following by four days of discontinuation, up to four cycles
  Interventions: Drug: Condylox Topical Gel 0.5%
- Placebo Gel (Placebo Comparator): Subjects in this arm will receive a vehicle that matches the test product, except for the inclusion of the active ingredient
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: Podofilox Gel 0.5% — Apply twice daily for three consecutive days, then discontinuing for four consecutive days, up to four treatment cycles
  Arms: Podofilox Gel 0.5 %
Drug: Condylox Topical Gel 0.5% — Apply twice daily for three consecutive days, then discontinuing for four consecutive days, up to four treatment cycles
  Arms: Condylox Topical Gel 0.5%
Drug: Placebo Gel — Apply twice daily for three consecutive days, then discontinuing for four consecutive days, up to four treatment cycles
  Arms: Placebo Gel

SUMMARY:
A clinical endpoint bioequivalence (BE) study for a Podofilox Gel 0.5% formulation for the treatment of external anogenital warts in comparison to Condylox® Gel 0.5% that follows the study design and recommendations according to Office of Generic Drugs (OGD) of U.S. Food and Drug Administration (FDA) Draft Guidance for Podofilox recommendations

DETAILED DESCRIPTION:
This is a multicenter, parallel group, randomized, double-blind, placebo-controlled, trial with clinical endpoint comparing Podofilox Topical Gel 0.5% to Condylox® Gel 0.5% and a matching placebo. The study will be conducted among adult male and female patients with external anogenital warts. The Investigator will assess vital signs and perform physical examination identifying any clinically significant abnormalities. Laboratory samples will be collected, including HIV, Hepatitis B&C, and urine pregnancy tests (UPT) for women of childbearing potential. The Investigator will confirm the diagnosis of External Anogenital Warts (EAW) and the absence of contraindications specified in the exclusion criterion 4 during the visual examination. The biopsy of skin lesions will be performed per the discretion of the Investigator for microscopic verification of the diagnosis of EAWs if any doubts of the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to participating in this study.
2. Male or female subjects, aged 18-65 inclusive, with a clinical diagnosis of external anogenital warts (i.e., perianal warts and/or external genital warts), including two or more distinct external genital warts, and wart area that is equal or less than 10 cm2. Histological confirmation should be obtained if there is any doubt of the diagnosis.
3. Females of childbearing potential may be enrolled if they practice a method of birth control with a reliability of at least 90%.
4. Sexually active study participants must agree to abstain from sexual activity of any kind throughout the treatment period to prevent cross- and reinfection by HPV.
5. Any female subject with childbearing potential has a negative urine pregnancy test at Baseline.
6. Negative HIV test within 4 weeks before Baseline.

   Exclusion Criteria:
7. Female subjects who are pregnant or lactating or planning to become pregnant during the study period.
8. Hypersensitivity or intolerance to Podofilox or any component of the formulation.
9. History of previous unsuccessful treatment with any formulation of Podofilox.
10. Wart area that is greater than 10 cm2.
11. Patients with internal anogenital and mucous membrane warts, Bowenoid papulosis, squamous cell carcinoma, active herpes lesion, or other skin abnormalities of treatment area, such as eczema, or skin that had not healed following surgery (cryosurgery, laser ablation or similar).
12. Primary or secondary immunodeficiency.
13. Known presence of diabetes type I or II.
14. Local irritation in any treatment area that would interfere with treatment.
15. Use within 4 weeks prior to baseline of any: 1) treatment for anogenital warts, 2) systemic corticosteroids, or 3) systemic immunosuppressive drug.
16. Any medical or surgical condition in the judgment of the Investigator that may interfere with the assessment of efficacy or safety, or pose a risk to the subject.
17. Patients known to abuse alcohol and/or drugs, or with a history of chronic alcohol or drug abuse that may result in protocol noncompliance.
18. Received another investigational drug, device or biologic within 90 days prior to the start of Screening or has planned to participate in another clinical trial while enrolled in this study.
19. Subjects who in the opinion of the investigator, are unlikely to be able to follow the restrictions of the protocol and complete the study
20. Employee (or employee's family member) of the research center or private practice, CRO or Sponsor, or subjects who have a conflict of interest.
21. Subjects living (e.g., siblings, spouses, relatives, roommates) in the same household cannot be enrolled in the study at the same time.
22. Previous enrollment in this study, current enrollment in this study at another participating site or current enrollment in another study (in parallel to this study) at another clinical research site.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evgeniy Cherepanov, MD, Study Director — bioRASI, LLC
Locations (17):
- United States (4):
  - Leon Medical Research, Miami, Florida
  - Well Pharma Medical Research Corp, Miami, Florida
  - Paddington Testing Co, Inc, Philadelphia, Pennsylvania
  - TMC Life Research, Inc, Houston, Texas
- Russia (8):
  - "Ecology of Health" LLC, Chelyabinsk
  - State Budgetary Institution of Healthcare "Chelyabinsk Regional Clinical Dermatovenerology Dispensary", Chelyabinsk
  - State autonoumous institution of Healthcare of Moscow region "Korolev Dermatovenerology dispensary", Korolyov
  - "Moscow scientific-practical center of Dermatovenerology and cosmetology", Moscow
  - "Clinic of urology №1" LLC, Penza
  - Rostov State Medical University, Rostov-on-Don
  - State Budgetary Institution of Healthcare "Dermatovenerologic dispensary #8" of Krasnogvardeyskiy district of Saint Petersburg, Saint Petersburg
  - Regional State-Financed Health Institution of Healthcare "Smolensk Dermatovenerologic dispensary", Smolensk
- Ukraine (5):
  - Medical Center of Private Enterprise "Dzerkalo", Dnipro
  - Municipal institution "Ivano-Frankivsk Regional Clinical Skin and Venereal Dispensary", Ivano-Frankivsk
  - Municipal Health Care Institution "Kharkiv City Clinical Dermatovenerologic Dispensary №5", Kharkiv
  - Municipal Institution "Rivne Regional Dermatology and Venerology Dispensary" of Rivne Regional Council, Rivne
  - Municipal Institution "Zaporizhzhya Regional Dermatovenerology Clinical Dispensary" of Zaporizhzhya Regional Council, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Podofilox Gel 0.5 % | Condylox Topical Gel 0.5% | Placebo Gel
Started | 201 | 198 | 67
Completed | 196 | 194 | 63
Not Completed | 5 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Podofilox Gel 0.5 % | Condylox Topical Gel 0.5% | Placebo Gel | Total
Number analyzed (Participants) | 201 | 198 | 67 | 466
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 201 | 198 | 67 | 466
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (12.745) | 37.7 (11.24) | 32.3 (10.401) | 34.7 (11.705)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 83 | 28 | 196
  Male | 116 | 115 | 39 | 270
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 38 | 17 | 91
  Not Hispanic or Latino | 165 | 160 | 50 | 375
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 19 | 14 | 5 | 38
  White | 176 | 180 | 62 | 418
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
  other | 4 | 4 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects With Total Disappearance of All Warts Within All Treated Areas.
Description: The primary endpoint is the Number and Percentage of subjects in the per protocol (PP) population with "treatment success" defined as "total disappearance of all warts within all treated areas".
Time Frame: 28 days.
Population: Due to GCP non-compliance in site 201, two sets of Efficacy Analysis were generated: Definitive Efficacy Analysis Set excluding site 201 and Supplemental Efficacy Analysis Set including site 201. Analysis using Definitive Efficacy Analysis Set (without site 201) were considered definitive for bioequivalence. The same analyses were performed using supplemental efficacy analysis set (sensitivity analysis) and these analyses were considered supportive.
Measure: Count of Participants; unit: Participants
Arm/Group | Podofilox Gel 0.5 % | Condylox Topical Gel 0.5% | Placebo Gel
Number analyzed (Participants) | 155 | 153 | 52
Participants | 100 | 102 | 12
Statistical Analysis 1: Comparison: Podofilox Gel 0.5 % vs Condylox Topical Gel 0.5%; Test type: Equivalence — BE limits: -20.0% to 20.0%; Equivalence ratio = 0.98, 90% CI 2-sided [-12 to 7]

2. Secondary Outcome: Local Application Site Reaction Scores (Erythema, Dryness, Burning/Stinging, Erosion, Edema, Pain, Itching, and Bleeding) Per Skin Reaction Scale.
Description: Local application site reactions scores (erythema, dryness, burning/stinging, erosion, edema, pain, itching and bleeding) in each group during the study drug application period. Other adverse events including serious adverse events throughout the study participation. Local skin reaction scores for erythema, dryness, burning/stinging, erosion, edema, pain, itching and bleeding will be recorded by the Investigator for every study visit based on their intensity. Skin Reaction Scale will be used absent, mild (slight, barely perceptible), moderate (distinct presence) and severe (marked, intense).
Time Frame: 28 days (at visit 6)
Population: Safety Population, 266 subjects completed the study at visit 6 (Podofilox Gel 0.5%: 114 subjects; Condylox Topical Gel 0.5%: 102 subjects and Placebo gel: 50 subjects).
Measure: Count of Participants; unit: Participants
Arm/Group | Podofilox Gel 0.5 % | Condylox Topical Gel 0.5% | Placebo Gel
Number analyzed (Participants) | 114 | 102 | 50
Participants
  Erythema: Absent | 102 | 81 | 45
  Erythema: Mild | 9 | 14 | 4
  Erythema: Moderate | 3 | 7 | 1
  Erythema: Severe | 0 | 0 | 0
  Dryness: Absent | 111 | 94 | 50
  Dryness: Mild | 3 | 7 | 0
  Dryness: Moderate | 0 | 1 | 0
  Dryness: Severe | 0 | 0 | 0
  Burning/Stinging: Absent | 108 | 92 | 48
  Burning/Stinging: Mild | 4 | 5 | 1
  Burning/Stinging: Moderate | 2 | 5 | 1
  Burning/Stinging: Severe | 0 | 0 | 0
  Erosion: Absent | 111 | 97 | 50
  Erosion: Mild | 1 | 2 | 0
  Erosion: Moderate | 2 | 3 | 0
  Erosion: Severe | 0 | 0 | 0
  Edema: Absent | 112 | 98 | 50
  Edema: Mild | 2 | 4 | 0
  Edema: Moderate | 0 | 0 | 0
  Edema: Severe | 0 | 0 | 0
  Pain: Absent | 114 | 99 | 50
  Pain: Mild | 0 | 3 | 0
  Pain: Moderate | 0 | 0 | 0
  Pain: Severe | 0 | 0 | 0
  Itching: Absent | 111 | 94 | 49
  Itching: Mild | 1 | 6 | 1
  Itching: Moderate | 2 | 2 | 0
  Itching: Severe | 0 | 0 | 0
  Bleeding: Absent | 114 | 102 | 50
  Bleeding: Mild | 0 | 0 | 0
  Bleeding: Moderate | 0 | 0 | 0
  Bleeding: Severe | 0 | 0 | 0

3. Secondary Outcome: Analysis of Safety Variables Will be Based on All Adverse Events (AE).
Description: AEs will be summarized based on the frequency of AEs and their severity for all treated subjects.
Time Frame: The AE reporting period for this study begins with the signature of the Informed Consent Form and, for unresolved AEs, ends 30 days following the last study medication application, a total of up to 65 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Podofilox Gel 0.5 % | Condylox Topical Gel 0.5% | Placebo Gel
Number analyzed (Participants) | 201 | 198 | 67
Participants
  Number of subjects with at least One TEAE | 105 | 114 | 33
  Number of Subjects with at Least One Related TEAE | 102 | 105 | 29
  Number of Subjects with at Least One Severe TEAE | 4 | 1 | 0
  Number of Subjects with at Least One TEAE Leading to Discontinuation | 1 | 1 | 0
  Number of Subjects with at Least One TEAE Leading to Death | 0 | 0 | 0
  Number of Subjects with at Least One TESAE | 0 | 1 | 0
  Number of Subjects with at Least One Related TESAE | 0 | 1 | 0
  Number of Subjects with at Least One Severe TESAE | 0 | 1 | 0
  Number of Subjects with at Least One TESAE Leading to Discontinuation | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: The AE reporting period for this study begins with the signature of the Informed Consent Form and, for unresolved AEs, ends 30 days following the last study medication application, a total of up to 65 days.
Arm/Group | Podofilox Gel 0.5 % | Condylox Topical Gel 0.5% | Placebo Gel
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/198 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/201 | 1/198 | 0/67
Other Adverse Events (participants affected / at risk) | 105/201 | 114/198 | 33/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Podofilox Gel 0.5 % (N=201) | Condylox Topical Gel 0.5% (N=198) | Placebo Gel (N=67)
Application Site Necrosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Podofilox Gel 0.5 % (N=201) | Condylox Topical Gel 0.5% (N=198) | Placebo Gel (N=67)
Application site erythema (General disorders) | 69 | 79 | 20
Application site pain (General disorders) | 52 | 56 | 16
Application site pruritus (General disorders) | 24 | 26 | 7
Application site dryness (General disorders) | 19 | 17 | 4
Application site erosion (General disorders) | 15 | 19 | 1
Application site erosion (General disorders) | 6 | 10 | 5
Application site haemorrhage (General disorders) | 2 | 2 | 0
Application site necrosis (General disorders) | 0 | 1 | 0
Feeling hot (General disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 2
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 3 | 2
Paraesthesia (Nervous system disorders) | 1 | 1 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyperaemia (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any use of information, data or results related to, associated with and directly resulting from the Study shall only be published or presented only after providing a copy of the manuscript or presentation, at least 60 days in advance of such publication or presentation, to the Sponsor for its review and approval in writing. No Confidential Information may be published without the express written consent of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT03532776/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT03532776/SAP_001.pdf